CLINICAL TRIAL: NCT01255605
Title: Impact of Intermittent Preventive Treatment (IPT) With Sulfadoxine-pyrimethamine (SP) on the Morbidities Associated With Malaria in Pregnant Women and Newborns in Peri-urban Areas of Bobo-Dioulasso, 5 Years After Its Adoption by the National Program for Fight Against Malaria in Burkina Faso.
Brief Title: Impact of IPT With Sulfadoxin Pyrimetamin on Pregnant Women and Their Babies Outcomes in Peri-urban Areas of Bobo-Dioulasso(Burkina Faso)
Status: Completed | Type: Observational
Sponsor: Université Polytechnique de Bobo-Dioulasso (Other)
Responsible Party: Principal Investigator, Dr Mamoudou Cisse, Medical doctor, Centre Muraz
Other Study IDs: PIC/INSSA/UPB-01
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Malaria, Pregnancy
Keywords: Intermittent preventive treatment with sulfadoxin-pyrimethamine; in Bobo-Dioulasso peri-urban areas, 5 years after its implementation; Burkina Faso.
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators make thick and thin blood smear and collect a few drops of blood on the 3MM paper Whatmann Schleicher-Schuell.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this is to determine the impact of intermittent preventive treatment (IPT) with sulfadoxine-pyrimethamine (SP) on the morbidities associated with malaria in pregnant women and newborns in rural peri-urban areas of Bobo-Dioulasso, 5 years after its implemented.

DETAILED DESCRIPTION:
Malaria in pregnant women is a crucial issue in Burkina Faso. Faced with this problem, a strategy based on the use of treated nets and intermittent preventive treatment (IPT) based on sulfadoxine-pyrimethamine (SP) was adopted in 2005. Five years after its implementation, the investigators will check whether this strategy is still effective in the preventing maternal and congenital malaria on the one hand and maternal anemia, low birth weight and prematurity on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the health area of Lafiabougou or secteur 24
* Having agreed to give free and informed consent

Exclusion Criteria:

* Bleeding from during the pregnancy
* eclampsia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our study population is constitued by pregnant women coming for antenatal care or delivery in two peripheral heath facilities of Bobo-Dioulasso(Lafiabougou and Secteur 24).
Sampling Method: Probability Sample
Enrollment: 772 (Actual)
Dates: Start 2010-09; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Peripheral and placental malaria | Peripheral malaria : at antenatal clinics and at delivery. Placental malaria: at delivery
  The investigators will check if pregnant women have any malaria parasites by making a finger prick thick respectively at antenatal clinics and at delivery. A placental thin smear will be made at delivery.

SECONDARY OUTCOMES:
Maternal anemia, congenital malaria,low birth weight, prematurity. | Maternal anemia: at antenatal clinics and at delivery. Congenital malaria: at delivery. Low birth weight: at delivery. Prematurity: at delivery.
  The investigators will check pregnant women haemoglobin level.A level< 11g/dl will be considered as anemia.
  Congenital malaria will be assessed through cord blood smear. Birth weight <2500g will be considered as low birth weight. Prematurity designs any birth before 37 gestation weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mamoudou Cisse, MD, Principal Investigator — Centre MURAZ Research Institute
Locations (1):
- Institut Supérieur des Sciences de la Santé/Université Polytechnique de Bobo-Dioulasso, Bobo-Dioulasso, Houet, Burkina Faso